CLINICAL TRIAL: NCT03864965
Title: Responses to a Standardized Approach to Advance Care Planning in Cognitive Disorders Clinic
Brief Title: Advance Care Planning in Cognitive Disorders Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201900108; ID00023545 (Other Grant/Funding Number: FL DOH); OCR21061 (Other: UF OnCore)
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Advance Care Planning
Keywords: Alzheimer's disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Advance Care Planning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients diagnosed with mild cognitive impairment, very mild dementia, or mild dementia, will receive the guided advance care planning conversations with the PI
  Interventions: Other: Advance Care Planning
- Control Patients (No Intervention): Patients diagnosed with mild cognitive impairment, very mild dementia, or mild dementia, will not receive the guided advance care planning conversations with the PI

INTERVENTIONS:
Other: Advance Care Planning — The provider will guide advance care planning conversations with patients identified with mild or moderate dementia during their third office visit, approximately three months after the first visit.
  Arms: Intervention Group

SUMMARY:
Advance care planning among patients with cognitive disorders poses unique challenges to clinicians. To improve planning in patients with Alzheimer's disease and other dementias, the researchers suggest a routine, standardized approach to these conversations. The main outcome measure is the rate of entry of Advance Directive completion in the patient's Electronic Health Record (EHR). A control group of similar patients from another provider specializing in cognitive disorders will be used to tease out confounding variable effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients having mild cognitive impairment (MCI) or very mild to mild dementia (CDR 0.5-1).

Exclusion Criteria:

* Patients with moderate to severe dementia (CDR 2-3).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Change in rate of advance directive completion during or following the visit | Baseline; Month 6; Month 12; Month 18
Change in the rate of completed advance directives that are uploaded to the patient's electronic medical record | Baseline; Month 6; Month 12; Month 18

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline; Month 2; Month 3
  Scale consisting of 14 items (7 relating to anxiety; 7 to depression). Scores range from 0-21 (0-7 being normal; 08-10 being borderline abnormal; 11-21 being abnormal for anxiety and depression).
Change in Beck Hopelessness Scale (BHS) | Baseline; Month 2; Month 3
  Scale consisting of 20 true-false items arrayed within three factors: Feelings about the future, loss of motivation, and future expectations. Scores range from 0-20 (0-3 as are considered within the normal range, 4-8 identify mild hopelessness, scores from 9-14 identify moderate hopelessness, and scores greater than 14 identify severe hopelessness).

CONTACTS AND LOCATIONS:
Overall Officials: Neal Weisbrod, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Department of Neurology, College of Medicine, UF Health Medical Plaza, Gainesville, Florida
  - UF Health Fixel Center for Neurological Diseases, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No